CLINICAL TRIAL: NCT05983770
Title: AT-1501-K207: BESTOW: A Phase 2, Multicenter, Randomized, Open-Label Study to Evaluate the Safety and Efficacy of Tegoprubart in Patients Undergoing Kidney Transplantation
Brief Title: Safety and Efficacy of Tegoprubart in Patients Undergoing Kidney Transplantation
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eledon Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AT-1501-K207; 2023-503336-41-00 (Other: European Clinical Trial Register); U1111-1278-5225 (Other: World Health Organization)
Record Dates: First submitted 2023-08-02; First posted 2023-08-09 (Actual); Last update posted 2025-10-29 (Actual); Status verified 2025-10

CONDITIONS: Kidney Transplant Rejection
Keywords: AT-1501; Kidney Transplant; Renal Allograft Rejection; Prophylaxis; CD40L Inhibitor; Humanized blocking antibody to CD40L; Monoclonal Antibody; Renal; Transplant; ESRD; Tegoprubart
MeSH Terms: conditions — Kidney Failure, Chronic | interventions — Tacrolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Investigative (Experimental): AT-1501 monoclonal antibody targeting CD40L given as an IV infusion
  Interventions: Drug: AT-1501
- Comparator (Active Comparator): Tacrolimus administered BID, targeting a whole blood trough concentration of 6-12 ng/mL until Month 6, and 6-8 ng/mL thereafter
  Interventions: Drug: Tacrolimus

INTERVENTIONS:
Drug: AT-1501 — IV infusions of AT-1501 20 mg/kg over 1 hour.
  Other Names: Tegoprubart
  Arms: Investigative
Drug: Tacrolimus — Tacrolimus will be administered BID, targeting a whole blood trough concentration of 6-12 ng/mL until Month 6, and 6-8 ng/mL thereafter.
  Arms: Comparator

SUMMARY:
This study will evaluate the safety and efficacy of AT-1501 compared with tacrolimus in patients undergoing kidney transplantation.

DETAILED DESCRIPTION:
This study is a randomized, multicenter, open-label, active control study to evaluate the safety and efficacy of AT-1501 compared with tacrolimus in the prevention of rejection in patients undergoing kidney transplantation. Up to 120 de novo kidney transplant recipients will receive rATG induction with corticosteroids (CS), and mycophenolate as maintenance therapy, and will be randomized 1:1 to receive either AT-1501 or tacrolimus.

ELIGIBILITY:
Inclusion Criteria:

* Male or female ≥ 18 years of age
* Recipient of their first kidney transplant from a living or deceased donor
* Agree to comply with contraception requirements during and for at least 90 days after the last administration of study drug

Exclusion Criteria:

* Induction therapy, other than study assigned rATG, planned as part of initial immunosuppressive regimen
* Currently treated with any systemic immunosuppressive regimen, including immunologic biologic therapies
* Currently treated with corticosteroids other than topical or inhaled corticosteroids
* Will receive a kidney with an anticipated cold ischemia time of > 30 hours
* Will receive a kidney from a donor that meets any of the following:

  * 5a. Donation after Cardiac Death (DCD) criteria; Or
  * 5b. Kidney Donor Profile Index (KDPI) of > 85%; Or
  * 5c. Is blood group (ABO) incompatible
* Medical conditions that require chronic use of systemic corticosteroids or other immunosuppressants
* History of a thromboembolic event, known hypercoagulable state, or condition requiring long term anticoagulation
* Positive T- or B-cell crossmatch that is due to HLA antibodies or presence of a DSA at Screening

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 127 (Actual)
Dates: Start 2023-08-30 (Actual); Primary Completion 2025-09-11 (Actual); Study Completion 2025-09-25 (Actual)

PRIMARY OUTCOMES:
eGFR at 12 months | Assessed from date of transplant through Day 364 (Month 12)
  Estimated Glomerular Filtration Rate (eGFR) at 12 months post-transplant

SECONDARY OUTCOMES:
NODAT at 12 months post-transplant | Assessed from date of transplant through Day 364 (Month 12
  The proportion of new onset diabetes after transplant (NODAT) at 12 months post-transplant
The proportion of patient and graft survival at 12 months post-transplant | Assessed from date of transplant through Day 364 (Month 12)
  Patient and graft survival are defined as either A) Death, B) re-transplantation or C) Requirement for regular dialysis
BPAR-free patient and graft survival at 12 months post-transplant | The proportion of BPAR-free patient and graft survival at 12 months post-transplant
  Assessed from date of transplant through Day 364 (Month 12)
BPAR at 12 months | Assessed from date of transplant through Day 364 (Month 12)
  The proportion of BPAR at 12 months

CONTACTS AND LOCATIONS:
Locations (43):
- United States (27):
  - University of California Los Angeles, Los Angeles, California
  - Keck School of Medicine of USC, Los Angeles, California
  - University of California, Irvine Medical Center, Orange, California
  - University of California, Davis Medical Center, Sacramento, California
  - Medstar Georgetown University Hospital, Washington D.C., District of Columbia
  - Tampa General Hospital, Tampa, Florida
  - Emory University Hospital, Atlanta, Georgia
  - Augusta University, Augusta, Georgia
  - University of Chicago, Chicago, Illinois
  - Loyola University Medical Center, Maywood, Illinois
  - University of Kansas Medical Center, Kansas City, Kansas
  - Tulane Medical Center, New Orleans, Louisiana
  - Johns Hopkins University, Baltimore, Maryland
  - Massachusetts General Hospita;, Boston, Massachusetts
  - Henry Ford Health System, Detroit, Michigan
  - University of Minnesota Medical Center, Minneapolis, Minnesota
  - Mayo Clinic, Rochester, Minnesota
  - Washington University in St. Louis, St Louis, Missouri
  - University of Nebraska Medical Center, Omaha, Nebraska
  - New York University Langone Health - Tisch Hospital, New York, New York
  - Duke University Medical Center, Durham, North Carolina
  - University of Cincinnati Medical Center, Cincinnati, Ohio
  - University of Pittsburgh Medical Center, Harrisburg, Pennsylvania
  - UT Southwestern, Dallas, Texas
  - Virginia Commonwealth University, Richmond, Virginia
  - University of Washington Medical Center, Seattle, Washington
  - University of Wisconsin Health, Madison, Wisconsin
- Australia (2):
  - Royal Adelaide Hospital, Adelaide, South Australia
  - Fiona Stanley Hospital, Perth, Western Australia
- Brazil (2):
  - Fundação Oswaldo Ramos - Hospital do Rim, São Paulo
  - Hospital das Clínicas da Faculdade de Medicina de São Paulo, São Paulo
- St. Paul's Hospital, Vancouver, British Columbia, Canada
- France (5):
  - Groupe Hospitalier Pellegrin, Bordeaux
  - CHU Grenoble-Alpes - Hopital Nord Michallon, Grenoble
  - Centre Hospitalier Universitaire Dupuytren, Limoges
  - CHU de Toulouse - Hopital de Rangueil, Toulouse
  - CHRU Tours - Hopital Bretonneau, Tours
- Charite Universitatsmedizin Berlin, Berlin, Germany
- Spain (5):
  - Hospital del Mar - Parc de Salut Mar, Barcelona
  - Hospital Universitari Vall d'Hebron, Barcelona
  - Hospital Clinic de Barcelona, Barcelona
  - Hospital Germans Trias i Pujol, Barcelona
  - Hospital Universitari de Bellvitge, Barcelona

IPD SHARING:
Plan to Share IPD: No